CLINICAL TRIAL: NCT04559750
Title: Internet Delivered Cognitive Behavior Therapy for Trichotillomania and Skin Picking Disorder
Brief Title: Internet CBT for Trichotillomania and Skin Picking Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Volen Ivanov, Principal Investigator, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-06325
Record Dates: First submitted 2020-09-08; First posted 2020-09-23 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-08

CONDITIONS: Trichotillomania; Excoriation (Skin-Picking) Disorder
MeSH Terms: conditions — Trichotillomania; Excoriation Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internet-delivered behavior therapy (I-BT (Experimental): 10 weeks of (I-BT) delivered via the Internet.
  Interventions: Behavioral: Internet delivered behavior therapy (I-BT)

INTERVENTIONS:
Behavioral: Internet delivered behavior therapy (I-BT) — 10 weeks of I-BT

SUMMARY:
The primary aim of the study is to test the feasibility, safety and efficacy of a manual based, Internet-delivered, behavior therapy (I-BT) for trichotillomania and skin picking disorder.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of trichotillomania and/or skin picking disorder according to DSM-5
* Living in Sweden with a Swedish personal identification number
* Able to participate in study assessment in Swedish and understand Swedish text
* Have regular access to a computer with Internet access and skills to use Internet
* Signed informed consent
* Outpatient

Exclusion Criteria:

* Psychotropic medication changes that can affect symptoms of trichotillomania or skin picking disorder within 2 months prior to treatment
* Other ongoing psychological treatments that could affect symptoms of trichotillomania or skin picking disorder
* Completed CBT for trichotillomania or skin picking disorder within the last 24 months
* Ongoing substance dependence or misuse
* Lifetime bipolar disorder or psychosis
* Suicidal ideation (a score of 5 points or higher on item 9 on the self-reported Montgomery-Åsberg depression rating scale
* Psychiatric comorbidity that could severely jeopardize treatment participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
The Massachusetts General Hospital Hairpulling Scale | Change from baseline (week 0) to post-treatment (week 10), 1-, 3-, 6- and 12-month follow-up.
  A self-report instrument for assessing repetitive hairpulling. The scale consists of seven items, rated for severity from 0 to 4 which assess urges to pull, actual pulling, perceived control, and associated distress.
The Skin Picking Scale - Revised | Change from baseline (week 0) to post-treatment (week 10), 1-, 3-, 6- and 12-month follow-up.
  A 6-item self-report measure of skin picking disorder severity.

SECONDARY OUTCOMES:
Montgomery Åsberg Depression Rating Scale Self Rate | Change from baseline (week 0) to post-treatment (week 10), 1-, 3-, 6- and 12-month follow-up.
  Total scores on the scale range from 0 to 54 with higher scores indicating a worse outcome (more severe depressive symptoms).
Sheehan Disability Scale | Change from baseline (week 0) to post-treatment (week 10), 1-, 3-, 6- and 12-month follow-up.
  Total scores on the scale range from 0 to 30 with higher scores indicating a worse outcome (higher degree of disability).
Acceptance and Action Questionnaire | Change from baseline (week 0) to post-treatment (week 10), 1-, 3-, 6- and 12-month follow-up.
  Total scores on the scale range from 10 to 70 with higher scores indicating a worse outcome (decreased levels of accpetance).
Acceptance and Action Questionnaire for Trichotillomania | Change from baseline (week 0) to post-treatment (week 10), 1-, 3-, 6- and 12-month follow-up.
  Total scores on the scale range from 9 to 63 with higher scores indicating a worse outcome (decreased levels of accpetance).
The Skin Picking Impact Scale | Change from baseline (week 0) to post-treatment (week 10), 1-, 3-, 6- and 12-month follow-up.
  Total scores on the scale range from 0 to 50 with higher scores indicating a worse outcome (higher impact of skin picking).
The NIMH Trichotillomania Symptom Severity Scale | Change from baseline (week 0) to post-treatment (week 10) and 12-month follow-up.
  Total scores on the scale range from 0 to 30 with higher scores indicating a worse outcome (higher symptom severity).
The NIMH Trichotillomania a Impairment Scale | Change from baseline (week 0) to post-treatment (week 10) and 12-month follow-up.
  Total scores on the scale range from 0 to 10 with higher scores indicating a worse outcome (higher impairment).
Patient Health Questionnaire 9. | Change from baseline (week 0) to post-treatment (week 10) and 12-month follow-up.
  Total scores on the scale range from 0 to 27 with higher scores indicating a worse outcome (more severe depressive symptoms).
EuroQol 5D, (EQ5D). | Change from baseline (week 0) to post-treatment (week 10) and 12-month follow-up.
  The responses of the individual are weighted and calculated from 1 (full health) to 0 (death). The measure also includes a self-rated health scale, which ranges from 0 to 100, with higher scores indicating better self-rated health.
Client Satisfaction Questionnaire-8. | Scores at post-treatment (week 10).
  Total scores range from 8 to 32, with higher scores indicating greater satisfaction with a health care service.
Treatment credibility scale. | Scores at mid-treatment (week 5) and post-treatment (week 10).
  The total score ranges from 1 to 10, with a higher score indicating a higher trust in the treatment.
Working Alliance Inventory - Short Form. | Scores at mid-treatment (week 5) and post-treatment (week 10).
  The scale ranges from 12 to 84, with higher scores indicating a stronger working alliance.
Clinical global impression - severity scale. | Change from baseline (week 0) to post-treatment (week 10)] and 12-month follow-up.
  Independent clinicians rate the severity of illness from "normal" (1) to "extremely ill" (7).
Clinical global impression - improvement scale. | Ratings at post-treatment (week 10) and at 12-month follow-up.
  Independent clinicians rate the improvement from "very much improved" (1), to "very much worse".
Global Assessment of functioning scale | Change from baseline (week 0) to post-treatment (week 10) and 12-month follow-up.
  Independent clinicians rate the symptoms and their effect on functioning from 1 to 100.
Negative events questionnaire (NEQ). | Ratings at post-treatment (week 10).
  The scale reports frequencies of negative events perceived by the participant as probably being caused by treatment and the negative impact of these events on a scale from 0 (not at all) to 4 (extreme).

CONTACTS AND LOCATIONS:
Locations (1):
- Psykiatri Nordväst, Stockholms Läns Sjukvårdsområde (SLSO), Region Stockholm, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No